CLINICAL TRIAL: NCT03314207
Title: Clinical Evaluation of Individuals With X-linked Retinitis Pigmentosa (XLRP) Caused by RPGR-ORF15 Mutations
Brief Title: Clinical Evaluation of Patients With X-linked Retinitis Pigmentosa (XLRP)
Status: Completed | Type: Observational
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AGTC-XLRP-001
Record Dates: First submitted 2017-10-11; First posted 2017-10-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP; retinal degeneration; RPGR; ORF15
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate subjects with X-linked retinitis pigmentosa caused by RPGR-ORF15 mutations in a clinical setting to fully characterize their condition, measure testing variability, and estimate rates of progression of clinical parameters.

DETAILED DESCRIPTION:
Males with a clinical diagnosis of X-linked retinitis pigmentosa (XLRP) caused by RPGR-ORF15 mutations will be asked to provide informed consent and will have a single blood or saliva sample obtained for DNA sequence analysis of genes known to cause XLRP, including the RPGR-ORF15 gene. All participants will be informed of the results of testing for these mutations. Those with qualifying mutations in the RPGR-ORF15 gene will be evaluated every 6 months for 3 years using a variety of non-invasive visual function tests to more fully characterize their clinical condition. Testing will include routine ophthalmic examinations and tests of visual acuity, perimetry, OCT, fundus imaging, and completion of quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with a clinical diagnosis of XLRP and a documented molecular diagnosis from a CLIA-certified laboratory of mutation within the ORF15 exon of the RPGR gene;
* At least 6 years of age;
* Willing and able to perform study procedures;
* Signed informed consent(s) obtained (and child assent where applicable).

Exclusion Criteria:

* Pre-existing eye conditions that would interfere with interpretation of study endpoints (e.g. glaucoma, corneal or lenticular opacities, diabetic retinopathy, history of retinal detachment);
* Participating in an interventional research study of drugs or devices for treatment of XLRP or other retinal diseases;
* Monoocular participants
* Any condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Males with a clinical diagnosis of X-linked Retinitis Pigmentosa (XLRP)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Disease progression in subjects with XLRP | Day 0 - Month 36

SECONDARY OUTCOMES:
Disease progression using visual acuity testing | Day 0 - Month 36
Disease progression using perimetry | Day 0 - Month 36
Disease progression using OCT | Day 0 - Month 36
Disease progression using electroretinography | Day 0 - Month 36
Disease progression using the National Eye Institute Visual Functioning Questionnaire-25 (VFQ-25) quality of life questionnaire | Day 0 - Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Feinsod, MD, Study Director — Applied Genetics Technologies Corporation
Locations (3):
- United States (3):
  - Duke Eye Center, Duke University Medical Center, Durham, North Carolina
  - Casey Eye Institute, Oregon Health and Sciences University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No